CLINICAL TRIAL: NCT04662840
Title: Prospective Blinded Study Looking at Geniculate Nerve Ablation of the Knee Versus Hyperemic Geniculate Artery Embolization Versus Sham Procedure for Pain Control in Patients With Knee Osteoarthritis
Brief Title: Geniculate Nerve Ablation vs Geniculate Artery Embolization vs Sham for Knee Osteoarthritic Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in getting participants to accept participating
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Louis-martin Boucher, Assistant professor/Staff Interventional Radiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-37-2021-6838
Record Dates: First submitted 2020-11-30; First posted 2020-12-10 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis, Knee
Keywords: artery embolization; nerve ablation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: three-arm prospective double-blinded randomized comparative trial
Who Masked: Participant, Care Provider
Masking Description: The referring surgeons, nursing staff, and the patient will all be blinded to outcome. Interventional radiologists and anesthetists performing the procedure itself cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham procedure (Sham Comparator): The patient will be placed on the procedural table as for the other arms. They will be blinded to what is occuring around them. A script detailing the procedure verbally will be followed by the interventionalists to "waste" time, but the only actual medical act that will be done is freezing of the skin around the knee (as for nerve ablation procedure) and at the groin (as for embolization procedure). Dressings will be applied at the knee and groin area.
  Interventions: Procedure: Skin infiltration of local anesthetic at groin and knee
- Geniculate artery embolization (Active Comparator): The patient will be placed on the procedural table as for the other arms. They will be blinded to what is occuring around them. They will undergo a similar script than everyone one else with freezing of the skin around the knee (as for the ablation procedure) and at the groin and in this group a geniculate artery embolization will be performed via an intraarterial access and use of embolization microspheres injected into the hypervascular arteries feeding the knee joint. Dressings will be applied at the knee and groin area.
  Interventions: Procedure: Geniculate artery embolization; Procedure: Skin infiltration of local anesthetic at groin and knee
- Geniculate nerve ablation (Active Comparator): The patient will be placed on the procedural table as for the other arms. They will be blinded to what is occuring around them. They will undergo a similar script than everyone one else with freezing of the skin around the knee and at the groin (as for the embolization procedure) and in this group a geniculate nerve ablation will be performed by advancing a radiofrequency ablation (RFA) needle at three locations alongside the tibia and femur where the nerves course and ablation performed. Dressings will be applied at the knee and groin area.
  Interventions: Procedure: Geniculate nerve ablation; Procedure: Skin infiltration of local anesthetic at groin and knee

INTERVENTIONS:
Procedure: Geniculate artery embolization — Under fluoroscopic guidance and angiographic imaging, a microcatheter is used to select all the arteries feeding the affected knee and Embosphere (100-300um) particles are injected to obtaining pruning of the hypervascular tissues arteries.
  Arms: Geniculate artery embolization
Procedure: Geniculate nerve ablation — Under fluoroscopic guidance, a Cool-tip RFA ablation needle is advanced such that it touches the femur at the condylar convexity on each side and the tibia at the tibial plateau convexity on the medial side. The ablation is performed to obtain an approximate zone of ablation of 2cm.
  Arms: Geniculate nerve ablation
Procedure: Skin infiltration of local anesthetic at groin and knee — Freezing of the skin will be performed at the groin (as prior to an arterial access for embolization procedure) and at three areas around the knee (as prior to insertion of the ablation needles for nerve ablation procedure).

SUMMARY:
This is a three-arm prospective double-blinded randomized comparative trial aimed at comparing results regarding knee pain improvement in patients with osteoarthritis (OA) of the knee awaiting total knee arthroplasty (TKA) by either a sham procedure, a geniculate artery embolization procedure or a geniculate nerve ablation procedure. Experienced interventional radiologists and anesthetists at the McGill University Health Centre (MUHC) and study affiliated centers will carry out all interventions. 72 consecutive subjects meeting the eligibility criteria, considered for knee replacement in the future. Patients will be randomized to receive either the embolization procedure, the nerve ablation procedure or a sham procedure. Monitoring of pain will be recorded using visual analog scales, pain medication use, and Western Ontario and McMaster Universities Arthritis Index (WOMAC) and osteoarthritis knee and hip quality of life questionnaire (OAKHQOL) questionnaires over a period of 1 year post-treatment or up to the time of surgery. Pain and recovery post surgery will be monitored as well in patients who do get the Total Knee Arthroplasty (TKA) before the 1 year mark.

DETAILED DESCRIPTION:
This is a three-arm prospective double-blinded randomized comparative trial. Experienced interventional radiologists and anesthetists at the MUHC and study affiliated centers will carry out all interventions.

* 72 consecutive subjects meeting the eligibility criteria, considered for knee replacement in the future.
* Patients will be referred for consideration for the study by specialized arthroplasty orthopedic surgeons from their osteoarthritis clinic at St-Mary's hospital.
* Prospective patients interested will be referred to the interventional radiology clinic at the MUHC for discussion of the procedures and of the study and recruitment.
* Consent will be obtained from all patients.
* Patients who accept to participate and fit the criteria will be randomized to receive either the embolization procedure, the nerve ablation procedure or a sham procedure. They will fill out the Western Ontario and McMaster Universities Arthritis Index (WOMAC) and osteoarthritis knee and hip quality of life questionnaire (OAKHQOL) questionnaires as well the Visual Analog Scale (VAS) for pain which will serve as baseline.
* They will then be contacted by the appropriate service to schedule the procedure.
* All embolization or nerve ablation procedures will be performed by either a qualified interventional radiologist or anesthetist.

Patients will be informed that they will not know which procedure they will receive. A barrier will be placed to shield them from visualizing the procedure and, for both procedures and sham procedure, skin freezing, and post-procedural bandages will be applied to the groin and in the skin around the knee. The patients will be informed that the procedures can take similar time between 15 minutes and 1 hr and that timing is variable between patients. They will also be informed that pain sensation around the knee can be similar between procedures. For all procedures, a written scenario (words and manipulations of the skin) will be followed such that all patients have the impression they are getting the same thing despite some having only the sham, others the embolization, and others the denervation. At the end of all procedures, patients will be transferred to the recovery room as per routine for interventional radiology procedures. Recovery room nurses will not know which of the procedures the patient had. They will be informed to look out for possible complications from either procedure. Patients will be informed that they must remain with their legs still for 3hrs after the procedure to prevent bleeding from the possible puncture in the artery that is necessary for the embolization procedure. No procedure specific technical discussion regarding the procedure will occur during the procedures to suggest what was done, only the common scenario will be followed. All this will be done in an attempt to blind the patient as much as possible. Blinding will be lifted for once the patient has completed the study. There is a final questionnaire to be filled out by the patient and physician at which point the patient will be informed of what procedure they received.

* The patients will be offered IV analgesia using midazolam and fentanyl during the procedure at regular intervals and the patients will be left to decide if they think it is necessary or not.
* Analgesics will be provided as per set orders during the recovery period in the post-procedural recovery room. Pain scales and medications provided are routinely registered in Post-Anesthesia Care Unit (PACU) documents and this data will be collected
* The patient will be discharged home with standard prescriptions for 2-3 days of post-procedural home analgesics and then will restart their routine pain control regimen they have been using.
* After the procedure, while at home, the patient will fill out paper or on-line confidential surveys (only study number on the survey, no patient identifying information) of routine medications used, WOMAC questionnaires and a VAS at regular interval (1d, 1wk, 2wks, 1m, 2m, 3m, 6m, 9m, 12m and if the patient has surgery at 1wk, 2wk, 1m, 2m, and 3m post-surgery). In addition, the OAKHQOL questionnaire will be filled out at 1m, 6m, and 12m and if the patient has surgery a 3m after surgery. The patients will be contacted by phone to make sure they remember to fill these out at the correct intervals. If they have chosen to use the paper forms, they will be collected in a pre-stamped envelope to send back to us at the 12m mark.
* A patient will be considered to have completed the study after 12m without knee surgery or 3m after a knee replacement surgery, whichever occurs first.
* Data will be gathered, stored, and analyzed.
* Data collected will include demographics, relevant medical history, vital signs, which procedure was performed, as well as the use of IV and oral analgesics, visual analog pain scores (VAS), WOMAC, and OAKHQOL questionnaires, X-rays performed during routine follow-ups at the orthopedic surgery clinic will be graded as per International Knee Documentation Committee (IKDC) grading system.
* Other than the initial visit aimed at getting consent and randomizing the patients and the procedures themselves, any research specific patient encounters scheduled in this study will be done by phone, unless the patient requests otherwise.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with knee osteoarthritis awaiting knee replacement surgery (expected to be more than a 3m waiting time) presenting with knee pain that patients consider unsatisfactorily managed by routine oral pain medications or cannot tolerate such medications.
2. Patients 18 y.o. or older

Exclusion Criteria:

1. Patients who are expected to have TKA surgery within 3 months.
2. Patients in whom the anatomy prevents either procedure

   * Vascular anatomy that prevents vascular access such as occluded vasculature to the leg
   * Skin or deep infection that would prevent placement of needles
3. Suspected concomitant infected knee joint or other signs of infections such as fever
4. Patients with uncorrectable abnormal coagulation status (INR >1.5 and plt < 50,000 without use of anticoagulation agents)
5. Patients who have known severe allergy to the anesthetic agent or contrast
6. Patients with pre-existing conditions, which, in the opinion of the investigator, interfere with the conduct of the study
7. Patients who are uncooperative, cannot follow instructions, or who are unlikely to comply with follow-up appointments or fill-out the post-procedural pain questionnaires
8. Patients with mental state that may preclude completion of the study procedure or be unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in knee pain post geniculate artery embolization versus nerve ablation vs sham | 1 year
  Assessment of changes in pain Visual Analog Scale (VAS - scale 0-10 with 10 being the highest degree of pain) scores between groups having undergone embolization versus ablation versus sham procedures
Changes in knee pain/functionality in geniculate artery embolization versus nerve ablation vs sham | 1 year
  Assessment of changes in pain and functionality score using Western Ontario and McMaster Universities Arthritis Index scores (WOMAC - scale 0-96 with 96 being the most worse pain/functionality) between groups having undergone embolization versus ablation versus sham procedures
Changes in pain medication use in geniculate artery embolization versus nerve ablation vs sham | 1 year
  Assessment in changes in dose (mg) of anti-inflammatory pain meds used between groups having undergone embolization versus ablation versus sham procedures

SECONDARY OUTCOMES:
Comparison of incidence of complications in geniculate artery embolization vs geniculate nerve ablation vs sham | 1 year
  Assessment of difference in incidence of serious complications (Grade C-E as per Society of Interventional Radiology (SIR) adverse event grading) in geniculate artery embolization vs geniculate nerve ablation vs sham groups
Changes in VAS pain scores after TKA in geniculate artery embolization vs geniculate nerve ablation vs sham | 3 months post-surgery
  Assessment of changes in pain (VAS - scale 0-10 with 10 being the highest degree of pain) scores post TKA between groups having undergone embolization vs geniculate ablation vs sham procedures
Changes in quality of life in geniculate artery embolization versus nerve ablation vs sham | 1 year
  Assessment of changes in functionality osteoarthritis knee and hip quality of life scores (OAKHQOL - scale 43 quality of life items scored from 0-10 with 10 being the worse symptoms) between groups having undergone embolization versus ablation versus sham procedures

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No